CLINICAL TRIAL: NCT04234087
Title: Feasibility and Effectiveness of an Additional Resistance and Balance Training in Cardiac Rehabilitation of Older Patients After Valve Surgery or Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Eglė Tamulevičiūtė-Prascienė, Head of a Rehabilitation department, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUHS001
Record Dates: First submitted 2020-01-12; First posted 2020-01-21 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Frailty Syndrome; Quality of Life; Valve Heart Disease
Keywords: Cardiac rehabilitation; Exercise training; Resistance training; Balance training; Physical capacity; Valve surgery; Valve intervention; Functional capacity
MeSH Terms: conditions — Frailty; Heart Valve Diseases | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The supervised exercise program included: continues endurance training on cycle ergometers (6 sessions a week). Every session included warm up (<50% target intensity 2 min, gradually increasing load 1-10 w/min up to target intensity within 5 - 10 min); exercise phase (100% of the target intensity (30-50% watts or 30-50% HRmax), starting with >5 minutes and gradually prolonged up to 30 min); cool down with gradual reduction of the load within 3 minutes); additional aerobic exercises performed sitting and/or standing (30 minutes, 5 days/week); respiratory muscle training (7 days/week, for 15 minutes) using ball trainer.
- Intervention group (Other): Exercise program as for a control group together with additional resistance and balance training 3 sessions/week. The resistance training was started with low intensity (<30% 1-RM, RPE ≤ 11, 5-10 repetitions), increased gradually to moderate intensity (30-50% and up to 60% 1-RM, RPE 12-13, after 8-15 repetitions) with 3 sets and 3 minute rest between sets, if tolerated. The balance training included exercises to improve static as well as dynamic balance ability. It was performed on 2-3 days/week for 10-15 minutes. The complexity of the balance exercises was selected and incremented individually by changing the stand-position, the base on which the stands were performed and/or using unstable surfaces. If tolerated, the visual information was varied and/or additional tasks performed while balancing. After completion participants were encouraged to continue exercise training at home according to recommendations.
  Interventions: Other: Additional balance and resistance training

INTERVENTIONS:
Other: Additional balance and resistance training — Additional exercise program with balance and resistance training three times per week. After completion participants are encouraged to continue exercise training at home according to recommendations and will receive control calls every two weeks.
  Arms: Intervention group

SUMMARY:
The aim of the study is to evaluate the short- and medium-term effectiveness of additional moderate dynamic resistance and balance training to the CR-program of old adults after valve surgery or intervention compared to usual care-CR.

ELIGIBILITY:
Inclusion Criteria:

* Patients after valve surgery and/or intervention
* Age 65 years and older
* Ability to start CR within 4 weeks after surgery,
* 6-minute walk distance (6-MWD) ≥100- ≤350 m (1)
* Patient's agreement to participate in the study.

Exclusion Criteria:

* Diseases in the musculoskeletal system or other organs complicating physical activity and exercise training;
* Exercise-limiting comorbidities (primarily orthopedic and neurological conditions that would exclude individuals from participating in CR according to study protocol), including chronic heart failure New York Heart Association Class IV, hemoglobin less than 9 g/dL, wound healing disturbance, cognitive or linguistic deficits.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 116 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Physical performance by Short Physical Perfromance Battery (SPPB) | Baseline
  The short physical performance battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests.The scores range from 0 (worst performance) to 12 (best performance).
Physical performance by Short Physical Perfromance Battery (SPPB) | 20 days
  The short physical performance battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests.The scores range from 0 (worst performance) to 12 (best performance).
Physical performance by Short Physical Perfromance Battery (SPPB) | Three months
  The short physical performance battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests.The scores range from 0 (worst performance) to 12 (best performance).
Physical performance by 5 meters walking test (5MWT) | Baseline
  5MWT is a gate speed test measured by meters per second.
Physical performance by 5 meters walking test (5MWT) | 20 days
  5MWT is a gate speed test measured by meters per second.
Physical performance by 5 meters walking test (5MWT) | 3 months
  5MWT is a gate speed test measured by meters per second.
Functional capacity by six minutes walking test (6MWT) | Baseline
  6MWT measured by meters
Functional capacity by six minutes walking test (6MWT) | 20 days
  6MWT measured by meters
Functional capacity by six minutes walking test (6MWT) | 3 months
  6MWT measured by meters
Quality of life by questionnaire Short Form Survey SF-36 | Baseline
  0-100%, the higher score, the better quality of life. The SF-36 measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH) in units on the scale
Quality of life by questionnaire Short Form Survey SF-36 | 20 days
  0-100%, the higher score, the better quality of life. The SF-36 measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH) in units on the scale
Quality of life by questionnaire Short Form Survey SF-36 | 3 months
  0-100%, the higher score, the better quality of life. The SF-36 measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH) in units on the scale
Quality of life by questionnaire Minnesota living with heart failure (Minesota HF) | Baseline
  Minesota HF questionnaire in units on the scale, 0-105, the the lower score, the better quality of life
Quality of life by questionnaire Minnesota living with heart failure (Minesota HF) | 20 days
  Minesota HF questionnaire in units on the scale, 0-105, the the lower score, the better quality of life
Quality of life by questionnaire Minnesota living with heart failure (Minesota HF) | 3 months
  Minesota HF questionnaire in units on the scale, 0-105, the the lower score, the better quality of life
Quality of life by questionnaire EQ-5D | Baseline
  EQ-5D in units on the scale, 0-10, the higher score, the better quality of life
Quality of life by questionnaire EQ-5D | 20 days
  EQ-5D in units on the scale, 0-10, the higher score, the better quality of life
Quality of life by questionnaire EQ-5D | 3 months
  EQ-5D in units on the scale, 0-10, the higher score, the better quality of life
Quality of life by questionnaire Quality of Life: Cardiac Index | Baseline
  Quality of Life: Cardiac Index in units on the scale, 15-33 the higher score, the better quality of life
Quality of life by questionnaire Quality of Life: Cardiac Index | 20 days
  Quality of Life: Cardiac Index in units on the scale, 15-33 the higher score, the better quality of life
Quality of life by questionnaire Quality of Life: Cardiac Index | 3 months
  Quality of Life: Cardiac Index in units on the scale, 15-33 the higher score, the better quality of life

SECONDARY OUTCOMES:
Frailty level by SPPB score | baseline
  Frailty measured by SPPB score - 0-7 - frail, 8-9 - pre-frail, 10-12 robust.
Frailty level by SPPB score | 20 days
  Frailty measured by SPPB score - 0-7 - frail, 8-9 - pre-frail, 10-12 robust.
Frailty level by SPPB score | three months
  Frailty measured by SPPB score - 0-7 - frail, 8-9 - pre-frail, 10-12 robust.
Frailty level by 5MWT | baseline
  Frailty measured by 5MWT - <0,6 m/s - frail, 0,7-0,99 m/s - pre-frail, 1,0 m/s and more - robust
Frailty level by 5MWT | 20 days
  Frailty measured by 5MWT - <0,6 m/s - frail, 0,7-0,99 m/s - pre-frail, 1,0 m/s and more - robust
Frailty level by 5MWT | three months
  Frailty measured by 5MWT - <0,6 m/s - frail, 0,7-0,99 m/s - pre-frail, 1,0 m/s and more - robust
Physical activity by International physical activity questionnaire (IPAQ) | 3 months
  IPAQ in units on the scale
Physical activity by International physical activity questionnaire (IPAQ) | 20 days
  IPAQ in units on the scale
Physical activity by International physical activity questionnaire (IPAQ) | Baseline
  IPAQ in units on the scale
Cardiopulmonary exercise capacity by maximal oxygen consumption (peakVO2) | Baseline
  PeakVO2 measured with spiroergometry by millilitres of oxygen per kilogram of body mass per minute
Cardiopulmonary exercise capacity by maximal load (maxWatt) | Baseline
  Maximal load measured with spiroergometry by maximal watts
Cardiopulmonary exercise capacity by maximal oxygen consumption (peakVO2) | 20 days
  PeakVO2 measured with spiroergometry by millilitres of oxygen per kilogram of body mass per minute
Cardiopulmonary exercise capacity by maximal oxygen consumption (peakVO2) | 3 months
  PeakVO2 measured with spiroergometry by millilitres of oxygen per kilogram of body mass per minute
Cardiopulmonary exercise capacity by maximal load (maxWatt) | 20 days
  Maximal load measured with spiroergometry by maximal watts
Cardiopulmonary exercise capacity by maximal load (maxWatt) | 3 months
  Maximal load measured with spiroergometry by maximal watts
Muscular strength by one repetition maximum test (1RM) | baseline
  1RM test for leg extension measured by kilograms
Muscular strength by one repetition maximum test (1RM) | 20 days
  1RM test for leg extension measured by kilograms
Muscular strength by one repetition maximum test (1RM) | 3 months
  1RM test for leg extension measured by kilograms

CONTACTS AND LOCATIONS:
Overall Officials: Raimondas Kubilius, Prof, Principal Investigator — Lithuanian University of Health Sciences, Department of Rehabilitation
Locations (1):
- LUHS hospital Kaunas Clinics Rehabilitation hospital of Kulautuva, Kaunas, Kulautuva, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tamuleviciute-Prasciene E, Beigiene A, Thompson MJ, Balne K, Kubilius R, Bjarnason-Wehrens B. The impact of additional resistance and balance training in exercise-based cardiac rehabilitation in older patients after valve surgery or intervention: randomized control trial. BMC Geriatr. 2021 Jan 7;21(1):23. doi: 10.1186/s12877-020-01964-3. PMID 33413144